CLINICAL TRIAL: NCT00979264
Title: Centers for Education on Research and Therapeutics - Heart Failure: Targeted Intervention Study
Acronym: CERTs-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00004022; 1U18HS016964 (AHRQ)
Record Dates: First submitted 2009-09-15; First posted 2009-09-17 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Heart Failure
Keywords: Quality Improvement
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Standard quality improvement approaches available through participation in Get With the Guidelines - Heart Failure.
- Intervention (Active Comparator): Enhanced and/or intensive quality improvement approaches, coupled with standard approaches available through participation in Get With the Guidelines - Heart Failure.
  Interventions: Behavioral: Intensive quality improvement tools

INTERVENTIONS:
Behavioral: Intensive quality improvement tools — Personalized performance improvement interventions, including premier site data reports, personalized feedback/teleconferences, comprehensive toolkits, and focused webinars; in addition to other general QI tools typically available through participation in Get With the Guidelines Heart Failure.
  Arms: Intervention

SUMMARY:
The objective of this study is to evaluate whether a quarterly feedback, education and performance improvement site-based intervention has a greater impact on quality performance and adherence to evidenced-based guidelines than existing on-demand feedback. This study will use a randomized design to compare changes in quality performance and adherence to selected measures among hospitals using existing on-demand reports and general quality improvement (QI) efforts versus those receiving intensive, targeted QI feedback via reports, teleconferences, webinars, and specialized tool kits.

ELIGIBILITY:
Inclusion Criteria:

* All sites participating in Get With the Guidelines Heart Failure.

Exclusion Criteria:

* Sites in Get With the Guidelines Heart Failure which opt out of participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Improvement in the overall opportunity-based composite of measures eligible for intervention (absolute score difference compared to the control arm) based on the existing Get With the Guidelines Heart Failure Achievement Measures and Quality Measures. | 1 year

SECONDARY OUTCOMES:
Improvement in Defect Free (all or none) score based on the combined Get With the Guidelines Heart Failure Achievement and Quality Measures | 1 year
Improvement in scores of each individual Get With the Guidelines Heart Failure Achievement and Quality Measure | 1 year
Improvement in length of stay and in-patient mortality. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eric D Peterson, MD, MPH, Principal Investigator — Duke Clinical Research Institute
Locations (1):
- Duke Clinical Research Institute, Durham, North Carolina, United States

REFERENCES:
- [Derived] DeVore AD, Cox M, Heidenreich PA, Fonarow GC, Yancy CW, Eapen ZJ, Peterson ED, Hernandez AF. Cluster-Randomized Trial of Personalized Site Performance Feedback in Get With The Guidelines-Heart Failure. Circ Cardiovasc Qual Outcomes. 2015 Jul;8(4):421-7. doi: 10.1161/CIRCOUTCOMES.114.001333. Epub 2015 Jul 14. PMID 26175533